CLINICAL TRIAL: NCT06564727
Title: Uniportal VATS Resection for Pulmonary Aspergilloma : Evaluation of Prognostic Factors in a Single Center Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hassan II University (Other)
Responsible Party: Principal Investigator, Sara WAGUAF, principal investigator, Hassan II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: pulmonary aspergilloma
Record Dates: First submitted 2024-08-14; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Pulmonary Aspergillosis; Surgery-Complications; Thoracic Diseases
MeSH Terms: conditions — Pulmonary Aspergillosis; Thoracic Diseases

STUDY DESIGN:
Intervention Model Description: study the effect of a treatment and evaluate outcome postoperatively
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uniportal VATS approach (Experimental): patient treated by Uniportal VATS technique
  Interventions: Procedure: Uniportal VATS approach
- VATS resection (Active Comparator): patients treated by VATS technique
  Interventions: Procedure: VATS approach

INTERVENTIONS:
Procedure: Uniportal VATS approach — Uniportal VATS resection for simple pulmonary aspergilloma
  Arms: Uniportal VATS approach
Procedure: VATS approach — VATS resection for complex pulmonary aspergilloma
  Arms: VATS resection

SUMMARY:
The objective of this study was to report our experience with U-VATS resection and to evaluate our surgical outcomes with an analysis of postoperative complications. The investigators also estimate the prognostic factors that influence the morbidity and the conversion.

DETAILED DESCRIPTION:
Evaluation of prognostic factors Tuberculosis Hemoptysis Type of aspergilloma presence of complete adherence Procedure

ELIGIBILITY:
Inclusion Criteria:

- Treatment using uniportal VATS

Exclusion Criteria:

- Resection using thoracotomy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
postoperative complications | 30 days
  evaluate the complication at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: sara WAGUAF, Principal Investigator — Hassan II University
Locations (1):
- Hassan II University, Casablanca, Morocco